CLINICAL TRIAL: NCT05565456
Title: Prospective Hounsfield Unit Measurements of Intercorporal Bone Grafts Remodelling Towards Spinal Fusion
Brief Title: Intercorporal Bone Graft Measurement Study
Status: Active, not recruiting | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NL81678.091.22; 2022-13716 (Other: METC Oost-Nederland)
Record Dates: First submitted 2022-09-27; First posted 2022-10-04 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Spondylolisthesis; Spinal Fusion
Keywords: Bone Density; Bone Remodelling; Tomography, X-Ray Computed
MeSH Terms: conditions — Spondylolisthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Instrumented lumbar fusion surgery is often accompanied by interbody fusion using an autologous bone graft that is supposed to expand and remodel to achieve a rigid and lasting bony construction between two vertebrae. However, there is a dearth of knowledge regarding the process of biological remodelling of intercorporal bone grafts. Also, a valid and reliable assessment of fusion status remains challenging because there is no objective tool available to quantify the bone remodelling process. CT-based Hounsfield Units correlate with Bone Mineral Density and can be used as a proxy to establish trajectories over time to assess changes in bone mineral density from the bone graft.

DETAILED DESCRIPTION:
Instrumented lumbar spinal fusion is a surgical procedure that is widely being used to treat various spinal diseases such as deformities, spondylolisthesis, spondylolysis, spinal instability, and degenerative disc disease. Lumbar fusion is an effective treatment to stabilize the degenerative segments and promote bony fusion and is often combined with subsequent decompression of neural structures or correction of deformities. To date, various surgical fusion techniques are used, but consensus regarding a superior technique is lacking. Also, the location where a surgeon wants to achieve bony fusion varies. Interbody fusion is performed to fuse the upper endplate of one vertebra and the lower endplate of the adjacent vertebra. An intervertebral cage is often used to retain intervertebral height and stability. After insertion of the cage, autologous decompressive bone is impacted behind the cage. Over time, this non-vital bone graft is expected to remodel towards new vital bone and subsequently to create a sustainable fusion between two adjacent lumbar vertebral bodies. However, in case of resorption of the bone graft or adequate bone remodeling, solid bridging of bone may fail to develop and this may result in a pseudarthrosis or non-union. This clinically important complication occurs in 5% to 35% of patients treated with spinal fusion and can lead to pain and a decrease in functional status. Also, subsequent revision surgery for symptomatic pseudarthrosis occurs in up to 24% of patients after fusion surgery.

The gold standard to assess interbody fusion is surgical exploration, but due to unpractical and ethical considerations, monitoring fusion status is mainly limited to radiographic image evaluation. CT-scanning is the most established radiographic method option for this, but when a patient improves clinically, conventional radiographs are used more commonly. An orthopaedic surgeon can use several existing scoring criteria to judge the degree of solid bony bridging based on this radiographic imaging. However, research has shown that the inter-observer agreement and diagnostic accuracy of these scoring criteria is relatively low. Correct diagnosis of lumbar fusion on CT has been reported to be as low as 67-72% and at the cervical level non-unions are missed in 20% of the cases. The problem is that, to date, there is no quantitative and objective tool available to quantify the bone remodeling process and to precisely judge whether vertebrae have fused or not. In fact, there is an overall dearth of knowledge about the biological process of ongoing spinal fusion and its association with the development of back and/or leg pain.

In vivo bone remodeling can be monitored by using repeated Bone Mineral Density (BMD) measurements. BMD values are traditionally generated using two-dimensional dual-energy X-ray absorptiometry (DEXA) scans which are hindered by overprojection from the iliac crest and metal artefacts. A more suitable proxy for these measurements is the use of Hounsfield Units (HU). HU can be measured on CT-images and highly correlate with BMD. HU have already been used to determine vertebral bone quality after spine surgery and have several clinical applications, including the ability to predict the stability of orthopaedic implants and to assist in surgical decision-making. However, none of these studies have succeeded in improving diagnostic accuracy in establishing spinal fusion.

Quantifying the biological bone remodeling process in the bone graft over time can help to evaluate bone growth or bone resorption. Knowledge of changes in bone mineral density from the bone graft could be very useful supplementary information when doubts about fusion status exist. To date, only two feasibility studies with relatively small sample sizes have reported on the value of HU measurements to evaluate bone graft remodeling after lumbar interbody fusion surgery. In one previous cross-sectional study from Spruit et al., published almost 18 years ago, HU measurements were only performed once in the first year after spinal fusion surgery. As such, no information with regards to the evolution of bone graft HU over time were obtained.

Recently the feasibility of HU measurements after lumbar spondylodesis (Reijmer et al, submitted) was explored. The HU measurement procedure that was developed during this study had excellent intraobserver reliability. The individual HU trajectories also suggested bone remodeling was not yet completed between one and two years after surgery. However, limitations of the study were a small sample size, the absence of postoperative CT-images made shortly after surgery and the absence of information about the participants' postoperative back and leg pain. This limited insight into the progression of pain and the process of bone graft remodeling in the first year after surgery. This study will build upon the results of the former study in an effort to further the state of the art in this important field of orthopaedics.

ELIGIBILITY:
Inclusion criteria:

* non-responsiveness to non-operative treatment in the six months prior to study enrolment
* fusion indicated for only one segment in the L1 to S1/ilium region
* between the age of 45 and 80.

Exclusion criteria:

* receiving revision spine surgery
* not wanting to provide informed consent
* pregnant or expecting to be pregnant within in the next two years.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty patients with a symptomatic spondylolisthesis (lytic/degenerative/iatrogenic) who have an indication for single level lumbar interbody fusion (PLIF/TLIF) will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Hounsfield Units (HU) | The HU will be assessed in the first week after surgery, at 6 months, at one year and at two years post-surgery.
  The participants' individual and group (mean, SD) HU values of their intercorporal bone graft(s) will be calculated from their (four) CT-scans.

SECONDARY OUTCOMES:
Intercorporal fusion | Intercorporal fusion will be assessed in the first week after surgery, at 6 months, at one year and at two years post-surgery.
  Intercorporal fusion will be assessed using the 5-point intercorporal fusion criteria by Brantigan et al.
Visual Analogue Scale (VAS) for back and leg pain. | Back and leg pain will be assessed at baseline, at 6 months, at one year and at two years post-surgery.
  Back and leg pain will be assessed using a (100mm) Visual Analogue Scale (VAS). A higher score indicates more pain.
Oswestry Low Back Pain Disability Questionnaire (ODI), Dutch version. | The degree of functional disability will be assessed at baseline, at 6 months, at one year and at two years post-surgery.
  The degree of functional disability will be assessed using the Dutch version of the Oswestry Low Back Pain Disability Questionnaire (ODI). Scores range from 0-50. A higher score (percentage) indicates a higher degree of functional disability.
36-item Research and Development (RAND-36) Health Survey, Dutch version. | The self-reported quality of life will be assessed at baseline, at 6 months, at one year and at two years post-surgery.
  The self-reported quality of life will be assessed using the Dutch version of the 36-item Research and Development (RAND-36) Health Survey. Scores range depending on the calculation method used. Higher scores indicate better self-reported quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Job LC van Susante, Dr. PhD., Principal Investigator — Rijnstate ziekenhuis
Locations (1):
- Rijnstate Hospital, Arnhem, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mobbs RJ, Phan K, Malham G, Seex K, Rao PJ. Lumbar interbody fusion: techniques, indications and comparison of interbody fusion options including PLIF, TLIF, MI-TLIF, OLIF/ATP, LLIF and ALIF. J Spine Surg. 2015 Dec;1(1):2-18. doi: 10.3978/j.issn.2414-469X.2015.10.05. PMID 27683674
- [Background] Cole CD, McCall TD, Schmidt MH, Dailey AT. Comparison of low back fusion techniques: transforaminal lumbar interbody fusion (TLIF) or posterior lumbar interbody fusion (PLIF) approaches. Curr Rev Musculoskelet Med. 2009 Jun;2(2):118-26. doi: 10.1007/s12178-009-9053-8. Epub 2009 Apr 29. PMID 19468868
- [Background] Chun DS, Baker KC, Hsu WK. Lumbar pseudarthrosis: a review of current diagnosis and treatment. Neurosurg Focus. 2015 Oct;39(4):E10. doi: 10.3171/2015.7.FOCUS15292. PMID 26424334
- [Background] Martin BI, Mirza SK, Comstock BA, Gray DT, Kreuter W, Deyo RA. Reoperation rates following lumbar spine surgery and the influence of spinal fusion procedures. Spine (Phila Pa 1976). 2007 Feb 1;32(3):382-7. doi: 10.1097/01.brs.0000254104.55716.46. PMID 17268274
- [Background] Fogel GR, Toohey JS, Neidre A, Brantigan JW. Fusion assessment of posterior lumbar interbody fusion using radiolucent cages: X-ray films and helical computed tomography scans compared with surgical exploration of fusion. Spine J. 2008 Jul-Aug;8(4):570-7. doi: 10.1016/j.spinee.2007.03.013. Epub 2007 May 29. PMID 17544854
- [Background] Kim KS, Yang TK, Lee JC. Radiological changes in the bone fusion site after posterior lumbar interbody fusion using carbon cages impacted with laminar bone chips: follow-up study over more than 4 years. Spine (Phila Pa 1976). 2005 Mar 15;30(6):655-60. doi: 10.1097/01.brs.0000155421.07796.7f. PMID 15770181
- [Background] Sakeb N, Ahsan K. Comparison of the early results of transforaminal lumbar interbody fusion and posterior lumbar interbody fusion in symptomatic lumbar instability. Indian J Orthop. 2013 May;47(3):255-63. doi: 10.4103/0019-5413.111484. PMID 23798756
- [Background] Williams AL, Gornet MF, Burkus JK. CT evaluation of lumbar interbody fusion: current concepts. AJNR Am J Neuroradiol. 2005 Sep;26(8):2057-66. No abstract available. PMID 16155160
- [Background] Brantigan JW, Steffee AD. A carbon fiber implant to aid interbody lumbar fusion. Two-year clinical results in the first 26 patients. Spine (Phila Pa 1976). 1993 Oct 15;18(14):2106-7. doi: 10.1097/00007632-199310001-00030. PMID 8272967
- [Background] Bridwell KH, Lenke LG, McEnery KW, Baldus C, Blanke K. Anterior fresh frozen structural allografts in the thoracic and lumbar spine. Do they work if combined with posterior fusion and instrumentation in adult patients with kyphosis or anterior column defects? Spine (Phila Pa 1976). 1995 Jun 15;20(12):1410-8. PMID 7676341
- [Background] Christensen FB, Laursen M, Gelineck J, Eiskjaer SP, Thomsen K, Bunger CE. Interobserver and intraobserver agreement of radiograph interpretation with and without pedicle screw implants: the need for a detailed classification system in posterolateral spinal fusion. Spine (Phila Pa 1976). 2001 Mar 1;26(5):538-43; discussion 543-4. doi: 10.1097/00007632-200103010-00018. PMID 11242382
- [Background] Soriano Sanchez JA, Soriano Solis S, Soto Garcia ME, Soriano Solis HA, Torres BYA, Romero Rangel JAI. Radiological diagnostic accuracy study comparing Lenke, Bridwell, BSF, and CT-HU fusion grading scales for minimally invasive lumbar interbody fusion spine surgery and its correlation to clinical outcome. Medicine (Baltimore). 2020 May 22;99(21):e19979. doi: 10.1097/MD.0000000000019979. PMID 32481262
- [Background] Brodsky AE, Kovalsky ES, Khalil MA. Correlation of radiologic assessment of lumbar spine fusions with surgical exploration. Spine (Phila Pa 1976). 1991 Jun;16(6 Suppl):S261-5. doi: 10.1097/00007632-199106001-00017. PMID 1862422
- [Background] Carreon LY, Glassman SD, Schwender JD, Subach BR, Gornet MF, Ohno S. Reliability and accuracy of fine-cut computed tomography scans to determine the status of anterior interbody fusions with metallic cages. Spine J. 2008 Nov-Dec;8(6):998-1002. doi: 10.1016/j.spinee.2007.12.004. Epub 2008 Feb 14. PMID 18280214
- [Background] van Bilsen MWT, Ullrich C, Ferraris L, Hempfing A, Hitzl W, Mayer M, Koller H. Diagnostic accuracy of CT scan-based criteria compared with surgical exploration for the analysis of cervical fusion and nonunion. J Neurosurg Spine. 2020 Mar 6;33(1):51-57. doi: 10.3171/2019.12.SPINE191011. Print 2020 Jul 1. PMID 32114527
- [Background] Schreiber JJ, Anderson PA, Hsu WK. Use of computed tomography for assessing bone mineral density. Neurosurg Focus. 2014;37(1):E4. doi: 10.3171/2014.5.FOCUS1483. PMID 24981903
- [Background] Lee S, Chung CK, Oh SH, Park SB. Correlation between Bone Mineral Density Measured by Dual-Energy X-Ray Absorptiometry and Hounsfield Units Measured by Diagnostic CT in Lumbar Spine. J Korean Neurosurg Soc. 2013 Nov;54(5):384-9. doi: 10.3340/jkns.2013.54.5.384. Epub 2013 Nov 30. PMID 24379944
- [Background] Demir O, Oksuz E, Deniz FE, Demir O. Assessing the effects of lumbar posterior stabilization and fusion to vertebral bone density in stabilized and adjacent segments by using Hounsfield unit. J Spine Surg. 2017 Dec;3(4):548-553. doi: 10.21037/jss.2017.09.05. PMID 29354730
- [Background] Schreiber JJ, Hughes AP, Taher F, Girardi FP. An association can be found between hounsfield units and success of lumbar spine fusion. HSS J. 2014 Feb;10(1):25-9. doi: 10.1007/s11420-013-9367-3. Epub 2013 Nov 1. PMID 24482618
- [Background] Nguyen HS, Shabani S, Patel M, Maiman D. Posterolateral lumbar fusion: Relationship between computed tomography Hounsfield units and symptomatic pseudoarthrosis. Surg Neurol Int. 2015 Nov 25;6(Suppl 24):S611-4. doi: 10.4103/2152-7806.170443. eCollection 2015. PMID 26693390
- [Background] Schreiber JJ, Anderson PA, Rosas HG, Buchholz AL, Au AG. Hounsfield units for assessing bone mineral density and strength: a tool for osteoporosis management. J Bone Joint Surg Am. 2011 Jun 1;93(11):1057-63. doi: 10.2106/JBJS.J.00160. PMID 21655899
- [Background] Spruit M, Meijers H, Obradov M, Anderson PG. CT density measurement of bone graft within an intervertebral lumbar cage: increase of hounsfield units as an indicator for increasing bone mineral content. J Spinal Disord Tech. 2004 Jun;17(3):232-5. doi: 10.1097/00024720-200406000-00011. PMID 15167340
- [Background] Reijmer JFH, de Jong LD, Kruyt MC, van Gorp MJ, Susante JLC. Repeated CT-based Hounsfield Unit Measurements as a Proxy Measure of Intercorporal Bone Graft Remodeling Towards Spinal Fusion; a Feasibility Study. [Submitted].

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT05565456/Prot_SAP_000.pdf